CLINICAL TRIAL: NCT00758537
Title: Tryptophan Metabolism in Kidney Disease
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. Petra Reinke MD, Charite UNiversity Medicine Berlin, Germany
Other Study IDs: TRY1STU
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Disease
Keywords: Assessment of tryptophan and tryptophan catabolites and IDO-activity in patients with chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (4):
- Patients with chronic kidney disease stage 3
- patients with chronic kidney disease stage 4
- patients with chronic kidney disease stage 5 (ESRD)
- Controls (no kidney disease)

SUMMARY:
Tryptophan metabolism in kidney disease will be investigated in patients with chronic kidney disease stages (ADOQI 3-5). Tryptophan levels and respective catabolites will be assessed under hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease (for > 3months) stages (National Kidney foundation/ADOQI): 3-5

Exclusion Criteria:

* Signs of infection or systemic inflammation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary care academic center, university hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-01; Study Completion 2008-10

PRIMARY OUTCOMES:
Course of plasma tryptophan level and levels of tryptophan metabolites under standard low-flux hemodialysis. | does not apply

CONTACTS AND LOCATIONS:
Overall Officials: Petra Reinke, Md PhD, Principal Investigator — Charite University Medicine
Locations (1):
- Charite University Medicine Berlin, Berlin, State of Berlin, Germany